CLINICAL TRIAL: NCT05971719
Title: Validation of a System Using Aerosol Glycerine to Detect and Localize Intraoperatively Pulmonary Air Leaks
Acronym: CT0136
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-11574
Record Dates: First submitted 2023-07-07; First posted 2023-08-02 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Air Leak From Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Air Leaks (Experimental): Lungs from patients undergoing lung transplantation after their removal from the recipient patient with previous informed consent signed before transplantation will be obtained. To establish a standard protocol to use our system we will use a dark box to validate that our system is able to localize the air leaks and to establish the best way to use the system. A one centimeter leak will be created on the lung with a scalpel. A laparoscope will be introduced via a trocar in the dark box and the surgeon will be asked to localize the leaks. The detection will be recorded via the laparoscope. The goal will be to perform a standardized protocol to use the system smoothly and efficiently on ex-vivo human lungs.
  Interventions: Diagnostic Test: Air Leaks: Aerosol glycerine System

INTERVENTIONS:
Diagnostic Test: Air Leaks: Aerosol glycerine System — A range of different leak will be done with different needle sizes on the lung. Perform localization on staple lines used surgically during pulmonary surgeries, as they are known to not consistently give an airtight closure. The lung will be put in the ex-vivo model and ask for a surgeon to localize the leaks with our system. The needle incisions will be repeat on another lung and ask the same surgeon to localize the leaks with the submersion test. To perform the submersion test the surgeon will have to submerge the lung in saline solution and to check the presence of air bubbles. The lung is inflated to pressures of 20 to 40 cm H209. The precision of both systems will be compared by the minimal incision the minimal incision the surgeon was able to localize.

SUMMARY:
Air leaks represent one of the most common complications and postoperative morbidity in thoracic surgery. Air leaks have been associated with the largest preventable morbidity associated with increased costs following lobectomy (typically related to increased length of stay). However, the standard used to detect and localize the air leaks, the submersion test, is not suitable for the standard surgical procedure, Video Assisted Thoracic Surgery. Considering the prevalence of this complication and the absence of a surgical standard of care for such complications, the aim of this study is to develop a system to create and send a glycerine aerosol smoke in the lungs of the patient. The smoke is visible with standard laparoscope and will flow though the pulmonary leak, thereby reducing postoperative surgical complications, morbidity, and length of stay for patients undergoing pulmonary resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lung transplant surgery
* Organ donor ineligible to donate lungs

Exclusion Criteria:

* Healthy individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Localization efficacy | 48 months
  Puncture the lungs to achieve an average size air leak (1-2 cm) and ask the surgeon to identify the airleak with the localization system. Register a success if the surgeon has properly localized the air leak and a failure if the surgeon has failed to localize the air leak. Destinguish the failures in false positive (Air leak detected in a non leaking area of the lung) and false negative (Air leak not detected when present). Compare that efficacy rate to the efficacy of a similar experiement done with the submersion technique.

SECONDARY OUTCOMES:
Duration of localization | 48 months
  Mesure the time required for the surgeon to localize the air leak area by the surgeon. Compare that time to the submertion test localization.
Minimal leak localizable | 48 months
  Puncture the lungs with different needle sizes and ask a surgeon to localize the air leaks on the lung. Record the smallest hole the surgeon was able to localize with our system. Then, compare the minimal leak localizable with our system to the minimal leak localizable with the submersion test.
Staple lines airtightness | 48 months
  Staple lines are known to not consistently give an airtight closure. But the manufacturers of those staple lines do not know why they are failing. Prove that the system can detect if the staple line is airtight or not, which could be useful for those manufacturers as well as for the clinicians. As leaks won't be created on every staple line, confirm that there is a leak by creating bubbles with saline at the staple line on the ex-vivo lung. Ask a surgeon to give the outcome of the airtightness of the staple line (success or failure) and then, compare the outcome to what we obtained with the localisation system.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUM, Montreal, Canada